CLINICAL TRIAL: NCT00000249
Title: Effects of Subanesthetic Concentrations of Nitrous Oxide
Brief Title: Effects of Subanesthetic Concentrations of Nitrous Oxide - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-08391-1; R01DA008391 (NIH); R01-08391-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Opioid-Related Disorders; Substance-Related Disorders
Keywords: nitrous oxide; subjective effects; healthy volunteer
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Control (No Intervention): Subject inhaled 0% N2O for 40 minutes with cold immersion at 10 and 30 minutes
- 20% N2O (Active Comparator): Subject inhaled 20% N2O for 40 minutes with cold immersion at 10 & 30 minutes
  Interventions: Drug: 20% N2O
- 30% N2O (Active Comparator): Subject inhaled 30% N2O for 40 minutes with cold immersion at 10 and 30 minutes
  Interventions: Drug: 30% N2O
- 40% N2O (Active Comparator): Subject inhaled 40% N2O for 40 minutes with cold immersion at 10 and 30 minutes
  Interventions: Drug: 40% N2O

INTERVENTIONS:
Drug: 20% N2O — 20% inhaled N2O
  Arms: 20% N2O
Drug: 30% N2O — 30% inhaled N2O
  Arms: 30% N2O
Drug: 40% N2O — 40% inhaled N2O
  Arms: 40% N2O

SUMMARY:
The purpose of this study is to conduct experiments to examine subjective and reinforcing effects of nitrous oxide. Mood altering and psychomotor effects will be tested on non-drug abusers and preference procedures will be used to assess reinforcing effects. To examine effects of subanesthetic concentrations of nitrous oxide on cold-pressor pain in humans.

ELIGIBILITY:
Please contact site for information.

Ages: 21 Years to 37 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 1993-09; Primary Completion 1995-06 (Actual); Study Completion 1995-06 (Actual)

PRIMARY OUTCOMES:
Pain intensity | during cold test at 10 min & 30 min of inhalation
  Subjects immersed non-dominant arm for 3 minutes twice in 2-3 degree C water while inhaling 0 (placebo), 20, 30, or 40% N2O for a total of 40 minutes

CONTACTS AND LOCATIONS:
Overall Officials: James Zacny, Ph.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Anesthesia & Critical Care, Chicago, Illinois, United States

REFERENCES:
- [Background] Pharmocol Biochem and Behavior 1995, 51( 2): 323-329